CLINICAL TRIAL: NCT05254717
Title: Effect of Soaking Complementary Foods Flour on Hemoglobin Concentration Level, Anthropometric Deficits and Episode of Diarrheal, Cough and Fever Morbidities of Children Age 6-24 Months
Brief Title: Effect of Soaking Complementary Foods Flour on Hemoglobin Concentration, Anthropometric Deficits and Episode of Diarrheal, Cough and Fever Morbidities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madda walabu university (Other)
Responsible Party: Principal Investigator, Mekonnen Tegegne, Principal Investigator, Madda walabu university
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MWU
Record Dates: First submitted 2022-02-02; First posted 2022-02-24 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Anemia
Keywords: Complementary feeding; soaking Flours; Undernutrition; Anemia
MeSH Terms: conditions — Anemia; Malnutrition | interventions — Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): Following baseline study, the interventional arm assigned to receive counselling intervention on complementary food flour soaking
  Interventions: Other: counselling
- control arm (No Intervention): The control group will be monitored for presence of any other intervention that might have a potential to mask the effect of the current intervention.

INTERVENTIONS:
Other: counselling — intervention groups will receive counselling on improving quality of complementary feeding by soaking complementary foods flours and basic methods of soaking complementary flours.
  Arms: Interventional arm

SUMMARY:
Removing anti nutrient factors using simple cost-effective and sustainable household methods to improve nutritional status of children in communities were plant based complementary foods are the main source of Nutrients is highly recommended. Therefore, the aim of this study is to determine effect of soaking complementary foods on hemoglobin, nutritional and health status of children 6-23 months in agrarian community of bale zone.

DETAILED DESCRIPTION:
Objectives of the intervention

* To determine prevalence and associated factors of nutritional status and anemia among children aged 6-23 months in agrarian community of Bale zone
* To Explore the complementary feeding practice knowledge perception of mother with children aged 6-23 months in agrarian community of Bale zone
* To determine effect of soaking complementary foods flour on nutritional status of children aged 6-23 months in agrarian community of Bale Zone
* To determine effect of soaking complementary foods flour on hemoglobin level of children aged 6-23 months in agrarian community of Bale Zone
* To determine effect of soaking complementary foods flour on frequency of morbidity of children aged 6-23 months in agrarian community of Bale Zone

Target groups The target groups for the intervention will be mothers with their children aged 6-23 months in selected Districts of Bale zone and participated in the baseline study.

Following baseline study, the two districts were assigned to be either an intervention or comparison group randomly. While the intervention community received the Nutrition counselling on promotion of complementary flour soaking, the comparison community was monitored for presence of any other intervention that might have a potential to mask the effect of the current intervention in the target. The intervention will be carried out for a period of six months.

End-line data collection included the following major components:

* Dietary Diversity practice
* Anthropometric measurements
* Hemoglobin test

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreed mothers with children aged 6-23 month

  * Mothers with children aged 6-23 month who lived at least six months in the selected communities
  * Mothers who have no plan to leave the area within 6 months period

Exclusion Criteria:

* • If the child is seriously ill at the time of data collection

  * Children with severe anemia hemoglobin level <= 7mg/dl will be excluded

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
children's blood hemoglobin concentration level | 15 days post intervention
children's Anthropometric deficits; Wasting (low-weight-for-length), stunting (low-Length-for-age) and underweight (low-weight-for-age) | 15 days post intervention
children's Episode of Diarrheal, cough and fever Morbidities | 15 days post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tefera Proff. Belachew, PHD, Study Director — Dean of School of Graduate Studies, Jimma University
Locations (1):
- Jimma University, Jimma, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tegegne M, Abate KH, Belechew T. Effect of counselling about complementary food flour soaking on nutritional and health status of children 6-23 months, a quasi-experimental study. Clin Nutr ESPEN. 2025 Apr;66:281-289. doi: 10.1016/j.clnesp.2025.01.038. Epub 2025 Jan 27. PMID 39864523